CLINICAL TRIAL: NCT07172282
Title: INFINITIVE: ImmuNotherapy For PatIeNts wIth colorecTal LIVer MEtastases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0340
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nelitolimod — Nelitolimod drug product is a clear to slightly opalescent, colorless to pale yellow solution free of visible particles and is supplied by TriSalus to the study sites in single-use vials. One vial is to be used per patient, and each vial should be discarded immediately after use.

SUMMARY:
Nelitolimod is a classC toll-like receptor 9 (TLR9) agonist that binds to TLR9 receptors on myeloid-derived suppressor cells(MDSCs) and helps reshape the tumor microenvironment (TME) and promote antitumor immunity. Investigators hypothesize that Nelitolimod can induce antitumor immune response in CRLM when administered regionally to the liver via a TriNav Pressure Enabled Drug Delivery (PEDD) catheter without compromising surgical feasibility or patient safety.

The study objective is to investigate the feasibility and safety of an innovative immunotherapeutic approach for patients with CRLM designed to overcome the immunosuppressive TME in CRLM. Investigators hypothesize that this investigational neoadjuvant treatment will be well tolerated and will not prevent patients from undergoing successful, safe CRLM liver resections. Investigators will assess the safety and feasibility of Nelitolimod given via TriNav PEDD in 10 patients with CRLM prior to liver resection. Patients will receive standard treatment with chemotherapy and then undergo placement of the PEDD catheter. Patients will then receive 3 doses of Nelitolimod before undergoing liver resection.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. A signed informed consent must be obtained prior to conducting any study-specific procedures.
* Male or female adults 18 years of age or older on day of signing informed consent.
* Radiographically confirmed metastatic adenocarcinoma to the liver from a colon or rectum primary tumor that is amenable to resection. TXNXM1+
* Only participants with liver-limited, resectable metastatic disease are eligible for participation (ablations are allowed to achieve an R0 intention-to-treat outcome).
* Only participants with pMMR (mismatch repair-proficient)/MSS mCRC are eligible. Microsatellite status should be performed according to the local standard of practice. (e.g., immunohistochemistry [IHC] and/or polymerase chain reaction [PCR], next-generation sequencing). Subjects with unknown or indeterminant results for either test at the time of enrollment are not eligible at investigators discretion.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1.
* Patients with synchronous disease who are planned to undergo liver and resection of primary are allowed.
* Total neoadjuvant therapy (TNT) for rectal cancers allowed.
* In the event the patient has had prior oxaliplatin-based adjuvant chemotherapy after resection of primary tumor, a minimum interval of 6 months should have passed prior to enrollment into the study.
* Patients must have completed standard of care FOLFOX/ FOLFIRI/FOLFIRINOX as part of pre- operative systemic therapy.
* Meets resectability criteria (all criteria MUST be met):

  1. Tumors that can be resected completely (R0), while leaving an adequate future liver remnant (defined under c.)
  2. The ability to preserve two contiguous hepatic segments with preservation of adequate vascular inflow and outflow as well as biliary drainage
  3. The ability to preserve adequate future liver remnant (>20 percent in a healthy liver; >30 percent after chemotherapy)
* Hematologic parameters defined as:

  1. Absolute neutrophil count (ANC) ≥ 1000 cells/mm3
  2. Platelet count ≥ 100,000/mm3
  3. Hemoglobin ≥ 8 g/dL
* Blood chemistry levels defined as:

  1. AST, ALT, alkaline phosphatase ≤5 times upper limit of normal (ULN)
  2. Total bilirubin ≤2x the ULN. Patients with Gilbert Syndrome should have a serum bilirubin ≤ 4x ULN and a direct bilirubin ≤2x ULN to be eligible.
* Adequate renal function as estimated by glomerular filtration rate (eGFR) >30 L/min determined based on the Cockcroft-Gault formula.
* Anticipated life expectancy greater than 6 months.
* Women of childbearing potential (WOCB) receiving systemic therapy should use effective contraception during treatment and for at least 9 months after the last investigational agent. Patients with partners who could become pregnant should use effective contraception during treatment and for 6 months after the last dose of investigational agent.

Exclusion Criteria:

* • Systemic therapy with immunosuppressive agents within 7 days or use of any investigational drug within 28 days before the start of trial treatment.

  * Prior exposure to any immune checkpoint blockade agent or any other immunomodulatory agent used as antineoplastic therapy for metastatic CRC.
  * Receipt of any organ transplantation, including allogeneic stem cell transplantation.
  * Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent, such as rheumatoid arthritis, which in the opinion of the Investigator might impair the subject's tolerance or ability to participate in the trial.
  * Known severe hypersensitivity reactions to monoclonal antibodies.
  * Failure to recover from any other toxicity (other than neuropathy or immune-related toxicity) related to previous anticancer treatment to grade ≤2.
  * Subject is pregnant or breast feeding or planning to become pregnant while enrolled in the study, up to the final (end of treatment) visit.
  * Participants unable to undergo endovascular placement of TriNav PEDD catheter due to any reason.
  * Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than 1 month before the start of study medication).
  * Congestive heart failure ≥ New York Heart Association (NYHA) class 2.
  * Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), myocardial infarction less than 6 months before start of study drug.
  * Uncontrolled cardiac arrhythmias.
  * Poorly controlled hypertension, defined as blood pressure consistently above 150/90 mmHg despite optimal medical management.
  * Major surgical procedure or significant traumatic injury within 28 days before start of study medication. Note: If participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
  * Non-healing wound, non-healing ulcer, or non-healing bone fracture.
  * Participants with evidence or history of any bleeding diathesis, irrespective of severity.
  * Any hemorrhage or bleeding event NCI CTCAE Grade ≥ 3 within 28 days prior to the start of study medication.
  * Significant acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease, malabsorption, or NCI CTCAE grade ≥ 2 diarrhea of any etiology.
  * Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus (T1DM), hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
  * Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
  * History of (non-infectious) pneumonitis that required steroids, current pneumonitis or interstitial lung disease.
  * Ongoing infection NCI-CTCAE grade >2 requiring systemic therapy.
  * Known history of positive test for HIV or known AIDS.
  * Any known positive test result for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating presence of virus, e.g. Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative).
  * Pregnant or lactating women.
  * Previous treatment with live vaccine within 30 days of planned start of study drugs (seasonal flu vaccines that do not contain a live virus are permitted).
  * Known history of allergy or hypersensitivity to study drug components.
  * History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial or interfere with the participation for the full duration of the trial.
  * Any condition that would prohibit the understanding or rendering of informed consent.
  * Any medical condition that in the opinion of the investigator would interfere with the patient's safety or compliance while on trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of neoadjuvant treatment with Nelitolimod delivered via PEDD in CRLM followed by surgical resection. | 24 months
  To assess the feasibility of neoadjuvant treatment with Nelitolimod delivered via PEDD in CRLM followed by surgical resection. Feasibility will be defined as at least 8 of 10 patients receiving surgery in a timely fashion (2-6 weeks). Enrollment will be stopped if 3 patients do not receive surgery in a timely fashion, irrespective of the number of patients enrolled. This is a safety and feasibility study for patients who as part of standard of care undergo liver resection.

SECONDARY OUTCOMES:
To assess the safety of Nelitolimod delivered via PEDD in CRLM. | 36 months
  To assess the safety of Nelitolimod delivered via PEDD in CRLM. To assess tumor regression score post-treatment with Nelitolimod and correlate with clinical outcomes, including: R0 rates, response (mRECIST), and DFS in resectable CRLM. AEs (graded by NCI CTCAE v5.0) attributed to the experimental drugs that prevent patients from getting the pre- planned surgery will be recorded, in addition to 30- day surgical complications rates. Tumor regression scores will be assessed post- treatment with Nelitolimod. The scores are based on a semiquantitative assessment of the ratio of viable tumor to fibrotic tissue. The scores range from 0 to 4, with 0 indicating no viable cancer cells and 4 indicating total regression. Tumor regression scores, response rate, and DFS are standard clinical parameters used to assess efficacy of a novel agent.

CONTACTS AND LOCATIONS:
Locations (1):
- RJ Zuckerberg, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No